CLINICAL TRIAL: NCT01282970
Title: Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Multiple Rising Oral Doses (5 to 100 mg q.d. for 14 Days) of BI 135585 XX in Patients With Type 2 Diabetes Mellitus (Randomized, Double-blind Placebo-controlled Within Dose Groups)
Brief Title: Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Multiple Rising Oral Doses of BI 135585 XX in Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1283.2; 2010-022698-32 (EudraCT Number: EudraCT)
Record Dates: First submitted 2011-01-24; First posted 2011-01-25 (Estimated); Last update posted 2014-11-19 (Estimated); Status verified 2014-11

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — 6-(2-hydroxy-2-methylpropyl)-3-(1-(4-(1-methyl-2-oxo-1,2-dihydropyridin-4-yl)phenyl)ethyl)-6-phenyl-1,3-oxazinan-2-one

ARMS (2):
- BI 135585 (Experimental): once daily doses as oral solution or tablet formulation over 14 days
  Interventions: Drug: BI 135585
- Placebo to BI 135585 (Placebo Comparator): once daily doses as oral solution or tablet formulation over 14 days
  Interventions: Drug: Placebo to BI 135585

INTERVENTIONS:
Drug: BI 135585 — oral doses given to approximately 5-6 parallel groups of 12 subjects (9 on active and 3 on placebo) over 14 days
  Arms: BI 135585
Drug: Placebo to BI 135585 — oral doses given to approximately 5-6 parallel groups of 12 subjects (9 on active and 3 on placebo) over 14 days
  Arms: Placebo to BI 135585

SUMMARY:
The objective of this study is to investigate safety, tolerability, pharmacokinetics and pharmacodynamics of BI 135585 XX following multiple dose administration over 14 days

ELIGIBILITY:
Inclusion criteria:

1. Male and postmenopausal or surgically sterilised female patients with an established diagnosis of type 2 diabetes mellitus prior to informed consent
2. Antidiabetic treatment with diet and exercise alone or with not more than one oral hypoglycaemic drug except glitazones, glucagon-like peptide 1 (GLP-1) analogues or dipeptidyl-peptidase 4 (DPP-4) inhibitors.
3. Antidiabetic treatment unchanged for 12 weeks prior to informed consent
4. Glycosylated haemoglobin A1 (HbA1c) ≤ 8.5% at screening
5. Age ≥ 20 and age ≤ 70 years
6. BMI ≥ 25 and BMI ≤ 40 kg/m2 (Body Mass Index)
7. Signed and dated written informed consent prior to admission to the study in accordance with GCP and the local legislation.

Exclusion criteria

1. Any finding of the medical examination (including BP, PR and ECG) deviating from normal and of not acceptable clinical relevance
2. Myocardial infarction, stroke or transient ischemic attack within 6 months prior to informed consent
3. Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders besides type 2 diabetes, hyperlipidaemia or medically treated hypertension
4. Gastrointestinal tract surgery that might affect absorption and elimination of drugs
5. Diseases of the central nerve system (such as epilepsy) or psychiatric disorders or relevant neurological disorders besides polyneuropathy
6. Chronic or relevant acute infections (e.g. HIV, hepatitis)
7. History of allergy/hypersensitivity (including allergy to drug or its excipients) that are deemed relevant to subject's safety or the trial by the investigator
8. Intake of drugs with a long half-life (> 24 hours) within one month prior to administration of the trial drug except for allowed co-medication
9. Treatment with glitazones, GLP-1 analogues, insulin, DPP-4 inhibitors, systemic or inhaled glucocorticoids, or anti-obesity drugs (e.g. orlistat) within 12 weeks prior to informed consent
10. Sensitive CYP3A4 substrates (e.g. simvastatin, lovastatin, verapamil, budesonide, buspirone, eplerenone , eletriptan, felodipine, fluticasone, midazolam, saquinavir, sildenafil, vardenafil) or CYP3A4 substrates with narrow therapeutic range (e.g. cyclosporine, ergotamine, pimozide, quinidine, sirolimus, tacrolimus, terfenadine) or drugs that prolong the QT/QTc interval (based on the knowledge at the time of protocol preparation) within 10 days prior to first administration of the trial drug
11. other exclusion criteria apply.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2011-02; Primary Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of BI 135585 will be assessed in a descriptive way using physical examinations (occurence of findings), vital signs, electrocardiograms, laboratory tests, and incidence and severity of adverse events. | up to 16 days post treatment

SECONDARY OUTCOMES:
Assessment of Pharmacokinetic parameter Cmax (maximum measured concentration of the analyte in plasma) of BI 135585 following single and multiple dose oral administration | up to 10 days post treatment
Assessment of Pharmacokinetic parameter tmax (time from dosing to maximum measured concentration) of BI 135585 following single and multiple dose oral administration | up to 10 days post treatment
Assessment of Pharmacokinetic parameter AUCτ,1 (area under the concentration-time curve of the analyte in plasma over a uniform dosing interval τ after administration of the first dose) | up to 10 days post treatment
Assessment of Pharmacokinetic parameter λz (terminal rate constant in plasma) of BI 135585 following single and multiple dose oral administration | up to 10 days post treatment
Assessment of Pharmacokinetic parameter Aet1-t2 (amount of analyte eliminated in urine from the time point t1 to time point t2) of BI 135585 following single and multiple dose oral administration | up to 10 days post treatment
Assessment of Pharmacokinetic parameter fet1-t2 (fraction of analyte eliminated in urine from time point t1 to time point t2) of BI 135585 following single and multiple dose oral administration | up to 10 days post treatment
Assessment of Pharmacokinetic parameter CLR,t1-t2 (renal clearance of the analyte from the time point t1 until the time point t2) of BI 135585 following single and multiple dose oral administration | up to 10 days post treatment
Assessment of Pharmacokinetic parameter Cmax,ss (maximum measured concentration of the analyte in plasma at steady state over a uniform dosing interval τ) of BI 135585 following single and multiple dose oral administration | up to 10 days post treatment
Assessment of Pharmacokinetic parameter tmax,ss (time from last dosing to maximum concentration of the analyte in plasma at steady state) of BI 135585 following single and multiple dose oral administration | up to 10 days post treatment
Assessment of Pharmacokinetic parameter Cpre,ss (predose concentration of the analyte in plasma at steady state immediately before administration of the next dose) of BI 135585 following single and multiple dose oral administration | up to 10 days post treatment
Assessment of Pharmacokinetic parameter AUCτ,ss (area under the concentration-time curve of the analyte in plasma at steady state over a uniform dosing interval τ) of BI 135585 following single and multiple dose oral administration | up to 10 days post treatment
Assessment of Pharmacokinetic parameter λz,ss (terminal rate constant in plasma at steady state) of BI 135585 following single and multiple dose oral administration | up to 10 days post treatment
Assessment of Pharmacokinetic parameter t1/2,ss (terminal half-life of the analyte in plasma at steady state) of BI 135585 following single and multiple dose oral administration | up to 10 days post treatment
Assessment of Pharmacokinetic parameter MRTpo,ss (mean residence time of the analyte in the body after multiple oral administrations at steady state) of BI 135585 following single and multiple dose oral administration | up to 10 days post treatment
Assessment of Pharmacokinetic parameter CL/F,ss (apparent clearance of the analyte in the plasma at steady state following extravascular multiple dose administration) of BI 135585 following single and multiple dose oral administration | up to 10 days post treatment
Assessment of Pharmacokinetic parameter Vz/F,ss (apparent volume of distribution during the terminal phase λz at steady state following extravascular administration) of BI 135585 following single and multiple dose oral administration | up to 10 days post treatment
Assessment of Pharmacokinetic parameter PTF (Peak-Trough Fluctuation) of BI 135585 following single and multiple dose oral administration | up to 10 days post treatment
Assessment of Pharmacokinetic parameter Cavg (average concentration of the analyte in plasma at steady state) of BI 135585 following single and multiple dose oral administration | up to 10 days post treatment
Assessment of Pharmacokinetic parameter Aet1-t2,ss (amount of analyte that is eliminated in urine at steady state from the time point t1 to time point t2) of BI 135585 following single and multiple dose oral administration | up to 10 days post treatment
Assessment of Pharmacokinetic parameter fet1-t2,ss (fraction of analyte eliminated in urine at steady state from time point t1 to time point t2) of BI 135585 following single and multiple dose oral administration | up to 10 days post treatment
Assessment of Pharmacokinetic parameter CLR,t1-t2,ss (renal clearance of the analyte in plasma from the time point t1 until the time point t2 at steady state) of BI 135585 following single and multiple dose oral administration | up to 10 days post treatment
Assessment of Pharmacokinetic parameter RA,Cmax (Accumulation ratio of the analyte in plasma at steady state after multiple dose oral administration over a uniform dosing interval τ, expresses ratio of Cmax at steady state and after single dose) | up to 10 days post treatment
Assessment of Pharmacokinetic parameter RA,AUC (Accumulation ratio of the analyte in plasma at steady state after multiple dose oral administration over a uniform dosing interval τ, expresses ratio of AUC at steady state and after single dose) | up to 10 days post treatment
Assessment of Pharmacokinetic parameter Cpre,N (the predose concentration of the analyte in plasma immediately before administration of the Nth dose after N-1 doses were administered) | up to 10 days post treatment
Exploratory evaluation of the pharmacodynamics of BI 135585 by determination of 11beta-hydroxysteroid dehydrogenase type 1 activity in adipose tissue (ex vivo) | up to 24 hours post treatment
Exploratory evaluation of the pharmacodynamics of BI 135585 by measuring of cortisol and cortisone and their metabolites in urine | up to 24 hours post treatment

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 1283.2.1 Boehringer Ingelheim Investigational Site, Neuss, Germany